CLINICAL TRIAL: NCT06709768
Title: Virtual Memory Attention and Problem Solving Skills for Persons With MS (MAPSS-MS) Pilot
Brief Title: Pilot of the Virtual Memory Attention and Problem Solving Skills Intervention for Persons With Multiple Sclerosis (MS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Alexa Stuifbergen, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY000066747
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis (MS)
Keywords: cognitive rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Individuals randomized to the intervention group will receive the MAPSS-MS virtually over an 8 week time period. The Virtual MAPSS-MS has two components: (1) group sessions via Microsoft teams with an expert facilitator focused on providing information and building efficacy for use of cognitive strategies, and (2) computer assisted cognitive training (Brain HQ).
  Interventions: Behavioral: Virtual Memory, Attention, and Problem Solving Skills for Persons with MS (MAPSS-MS)
- Wait List Control (No Intervention): Participants in this arm will complete data collection at the same time and intervals as the experimental arm. When all three data collections have been completed, they will be offered the opportunity to participate in the intervention - no additional data will be collected following the intervention.

INTERVENTIONS:
Behavioral: Virtual Memory, Attention, and Problem Solving Skills for Persons with MS (MAPSS-MS) — This is a pilot test of the MAPSS-MS intervention in a virtual delivery format.
  Arms: Intervention Group

SUMMARY:
The goal of this pilot clinical trial is to study is to test the feasibility and effects of a virtual (remote) version of a cognitive rehabilitation intervention - Memory, Attention, and Problem Solving Skills for Persons with MS (MAPSS-MS). We have already tested this intervention "in person" and found it to be effective at helping persons with MS improve their cognitive function learn. We are now testing the MAPSS-MS intervention using a virtual or remote format. The main questions this pilot study aims to answer are:

1. What is the feasibility of the Virtual MAPSS-MS intervention
2. Compared with persons in the wait list control group, will persons receiving the Virtual MAPSS-MS intervention have better overall neurocognitive function and 3. ) Compared with persons in the wait list control group, will persons receiving the Virtual MAPSS-MS intervention have improved stress, self-efficacy for cognitive everyday tasks, use of compensatory strategies and improved depressive symptoms, fatigue, sleep and pain.

Participants will be asked to take part in the MAPSS-MS intervention virtually and complete surveys and cognitive tests online at three time points: before the eight-week intervention, immediately after the intervention and six-weeks after the intervention.

The virtual MAPSS-MS has two components (a) Group sessions via zoom with an expert leader and (b) a computer assisted brain games (Brain HQ) program. The eight online group sessions (2 hours once per week) will address common cognitive concerns experienced by persons with MS and strategies that may be helpful. Participants will also be provided access to Brain HQ, a computerized training program, and asked to practice these games for 20-30 minutes on 5 or 6 days per week.

DETAILED DESCRIPTION:
This pilot study will use a randomized control trial experimental design with a wait list control group. Following completion of screening, consent and baseline data collection, participants will be randomized to either the Virtual MAPSSS intervention group or a wait list control. The intervention group will then receive the 8-week intervention via micorsoft teams and have access to Brain HQ to practice cognitive brain games. Both groups will complete Time 2 testing immediately after the 8-week intervention and Time 3 testing at 6 weeks following the intervention. Following all three data collection periods, the members of the wait list control will be offered the 8-week intervention if they wish to participate.

Recruitment and Screening procedures:

Recruitment will begin once approval is received from UT IRB. Participants may be recruited in a variety of ways including flyers in offices of physicians and service providers, targeted announcements to persons with MS on MS-Related web sites, contact with support groups, notices in MS newsletters and "word of mouth." Initially, we will contact individuals who indicated an interest in previous "in person" studies of the MAPSS-MS who were unable to participate due to difficulties with transportation, time, or distance. Furthermore, if needed, information about the study will be circulated on social media (Facebook and Instagram) and listed on the National Multiple Sclerosis Societies (NMSS) website. For the social media posts, the approved flyer will be posted from the research teams personal accounts. Group moderators for MS Support groups, who have a social media presence, will be contacted for permission to post our flyer and recruit in their group. All stated recruitment efforts will target local, regional, and national participants.

Potential participants who contact the research team will be screened for eligibility (as defined by the inclusion and exclusion criteria) via the telephone or via Microsoft Teams or Zoom by the study staff. The project staff will have a script to screen potential participants for inclusion/exclusion criteria and will explain the study procedures and requirements to those who are eligible. This will include administering the Perceived Deficits Questionnaire (Sullivan, Edgley & Dehoux, 1990) and asking questions regarding inclusion/exclusion criteria. Those with scores on the Perceived Deficits Questionnaire indicating they experience at least 5 problems "sometimes" or more often will be eligible to participate Since this data will only be used for recruitment purposes, only verbal consent will be obtained. If participants meet the criteria for the study over the phone, they will be invited for a one-on-one meeting when sufficient participants have been recruited to schedule the group sessions. The one-on-one meeting will include confirming the inclusion/exclusion criteria and a careful review of the informed consent. Participants that do not meet criteria at screening will be excluded and will be provided with information about the National MS Society website.

Participants who complete the screening will complete the baseline data (within 2 weeks of initiation of the intervention) and then be randomized to either the intervention or a wait-list control group, using a computerized table of random numbers.

Intervention Description. The overall purpose of the Virtual MAPSS-MS intervention is to help the individual acquire the highest level of cognitive functioning and functional independence. This is accomplished through teaching the use of compensatory skills, retraining skills (the computer games component) and environmental/lifestyle support for cognitive functioning. The Virtual MAPSS-MS has two components: (a) Group sessions via zoom with an expert facilitator focused on providing information and building efficacy for use of cognitive strategies and (b) an innovative computer-assisted cognitive rehabilitation (Brain HQ) program. The home-based computer component will enable the participants to engage in intensive practice sessions without leaving their homes. Translation of skills practiced to everyday issues will be a focus of the group sessions.

Group Component The investigators' prior work will drive the content and process aspects of the Virtual MAPSS-MS (Memory, Attention & Problem-Solving Skills for Persons with MS) intervention - specifically the health promotion intervention for women with MS (R01HD35047) and the multi-site trial of the 'in person' MAPSS-MS (1R01NR014362). The intent of the efficacy-based wellness intervention is to engage individuals in assessing their present health behaviors, setting meaningful goals for change and addressing the barriers, resources and skills necessary to improve health behaviors and consequently quality of life. In this study, we will use the same process and strategies (Stuifbergen, et al.,2012; Stuifbergen et al., 2018) to assist participants to acquire knowledge regarding the specific MS-related cognitive impairments; assess and acknowledge their cognitive concerns, build the skills necessary to implement compensatory self-management strategies of cognitive difficulties and set goals for integrating new cognitive skills into their everyday lives.

The group program will consist of weekly 2-hour online classes via Microsoft teams over an 8-week period with a trained facilitator who will present information, guide participants in self-assessment of cognitive problems, resources and barriers to cognitive functioning and enhancing self-efficacy for use of strategies to maximize cognitive functioning. Major topic areas will include (1) Identifying common cognitive problems experienced with MS (2) Compensatory Strategies to Maximize Cognitive Skills (3) Maximizing Cognitive Health with a MS - Lifestyle adjustments (e.g. physical activity and energy conservation) to promote cognitive functioning (4) Adjusting to Changes in Cognitive Skills (5) Stress Management (controlling anxiety) and Enhancing Cognition. At each session, the professional facilitator will evaluate the participants on Brain HQ exercises prescribed at the last session, troubleshoot cognitive strategies and performance difficulties, and prescribe the therapy exercise assignments for the upcoming week.

Computer Training Component (Brain HQ). The computer-training component, developed by Posit Science, uses a model for cognitive training that adapts to the user through an integrated hierarchical structure. The Brain HQ website houses the interactive program that runs on standard web browsers. Participants will only need a computer, smart phone, or tablet with Internet access to securely log onto the website. Each participant will be registered by the research staff using anonymous ID numbers that will allow unlimited access during the study. Participants will be provided with a unique email and password for the Brain HQ site and participant identifying information will not be used or submitted to Brain HQ. Staff will maintain a list of the assigned email and passwords so they can assist participants if needed. At the week 1 class, the interventionist will show participants how to log on and access the exercises via a screenshare option provided by the webinar program. The website stores each session a participant completes, and participants will be able to start subsequent sessions wherever they stopped the last time logged on. BrainHQ meets the Institute of Medicine's five requirements for a brain-training program: (1) transferability to other tested tasks; (2) transferability to real-world tasks; (3) evaluation with active control group with access to same product; (4) retention of trained skills; and (5) replication of findings. The intervention group will be asked to practice 20-30 minutes, 5-6 days a week. Study staff will be available via email to assist participants if they are having difficulty using the Brain HQ site.

Comparison Group. Those randomized to the wait list control group will complete all data collection at the same time intervals as those in the intervention group. When individuals have completed the 3rd data collection, they will be invited to participate in the MAPSS-MS zoom sessions over 8 weeks and be provided with access to the Brain HQ for home computer training. No additional data will be collected from the wait-list control group during this time period.

Data Collection. Questionnaire data will be collected from all participants via a secure link to REDCap at baseline (week 0), at completion of the intervention (week 8), and at 6 weeks post-intervention (week 14). Participants will also receive a separate email with a personalized link from the study coordinator to complete the neurocognitive test battery from CNS Vital Signs . The total data collection time will be about 60-70 minutes. Participants will receive a small incentive ($25) for completing the first two data collections and ($50) for the final assessment ($100 total). Data will be downloaded for analysis into SPSS.

ELIGIBILITY:
Inclusion Criteria: Age 21 -85 years old, reside in the United States, MS diagnosis for at least 1 years, access and ability to use phone, computer and Internet, Score of ≥10 on the Perceived Deficits Questionnaire (PDQ), adequate vision and motor skills to use the computer for testing and to participate in the intervention.

Exclusion Criteria:A diagnosis of dementia/head injury, inability to speak English, severe functional limitation that makes use of computer for intervention and testing impossible; prior participation in a cognitive rehab intervention during the last year; currently using Brain HQ at home.

-

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Function -Objective | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The Neurocognitive Index (NCI) score will be obtained via remote administration of the CNS Vital Sign's (CNS Vital Signs, LLC) Core computerized neurocognitive test battery. Batteries will be administered on participant's own computers. The core battery includes seven tests for verbal and visual memory, reaction time, processing speed, executive function, simple attention and motor speed, and five domain scores for composite memory, psychomotor speed, reaction time, cognitive flexibility, and complex attention The Neurocognitive Index is the average of five domain scores, representing a global score of neurocognition.
Perceived Cognitive Function PROMIS v2.0 - Cognitive Function-Abilities Short Form 8a | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The PROMIS v2.0 - Cognitive Function-Abilities Short Form 8a includes 8 items that assess patient-perceived cognitive deficits including the areas of mental acuity, concentration, verbal and nonverbal memory, and verbal fluency.

SECONDARY OUTCOMES:
Self-Efficacy for Cognitive Tasks | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The Self-Efficacy for Cognitive Everyday Tasks - Part IV consists of 25 items; that assess beliefs regarding one's ability to recognize, monitor and manage cognitive everyday cognitive activities (e.g. paying bills, recalling a list, planning).
Depressive Symptoms - CES-D 10 | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The CES-D - Short Form includes 10 item that measure the frequency of depressive symptoms during last 7 days. There is a 4-point item response scale from rarely/none of the time to most/all of the time.Higher scores indicate more frequent depressive symptoms.
Compensatory Strategies | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The Strategies to Improve Cognitive Function is a 20 item scale that assesses the use of compensatory strategies in everyday life. Higher scores indicate greater use of strategies.
Perceived Stress | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The Perceived Stress Scale includes 10 items that measure inidivual's perception of stress during the last month related to everyday challenges and life. Higher scores indicate greater perceived stress.
Pain Symptoms | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The PROMIS Pain Interference Short Form 4a will be used to measure the extent that pain has interfered with daily life during the last 7 days. Higher scores on the sum of the 4 item scale indicates greater pain interference.
Fatigue | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The PROMIS Fatigue Short Form 4 am will be used to measure the extent of overall fatigue and how fatigue affects life activities. The 4 items are summed and higher scores indicate greater fatigue.
Sleep | This measure will be completed at baseline, following the 8 week intervention and 6 weeks after the intervention is complete.
  The PROMIS Sleep Interference Form 4a is used to measure overall sleep quality and sleep disturbance in the last 7 days. Higher scores indicate greater disturbance of sleep.

IPD SHARING:
Plan to Share IPD: Yes
Other investigators may contact the PI for sharing of de-identified data.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from January 2026 to December 2028
Access Criteria: Individuals with PI status at other educational or research institutions may contact the study PI regarding data sharing. Specific plans will be developed in conjunction with the IRB that has study oversight.